CLINICAL TRIAL: NCT04316663
Title: Well-being Promotion and Sleep Hygiene Education to Improve Sleep Quality in a Non-clinical Population of Distressed Adults Reporting Poor Sleep: A Pilot Parallel-arm, Randomized Controlled Trial
Brief Title: Well-being Promotion and Sleep Hygiene Education to Improve Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Associate Professor of Nutritional Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAS8486
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Poor Quality Sleep
Keywords: Sleep Quality; Psychological Distress; Psychological Well-Being; Well-Being Therapy; Sleep Hygiene
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being; Sleep Hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Well-Being and Sleep Hygiene (Experimental): Participants in the experimental group will receive an intervention focused on both principles of psychological well-being and sleep hygiene education.
  Interventions: Behavioral: Well-Being Intervention; Behavioral: Sleep Hygiene
- Sleep Hygiene (Control) (Active Comparator): Participants in the control group will receive sleep hygiene education alone.
  Interventions: Behavioral: Sleep Hygiene

INTERVENTIONS:
Behavioral: Well-Being Intervention — The main aim of the well-being intervention is to reduce levels of distress through the promotion of psychological well-being. Key components of the intervention are self-monitoring of instances of well-being and what leads to their interruption (i.e., thoughts and behaviors), cognitive restructuring of interfering thoughts, and homework assignments to address dysfunctional behaviors and increase exposure to optimal experiences. Participants will become aware of their functioning based on six different dimensions of psychological well-being (i.e., self-acceptance, positive relations with others, autonomy, environmental mastery, purpose in life, and personal growth), and will be guided in finding a balance within each dimension.
  Arms: Well-Being and Sleep Hygiene
Behavioral: Sleep Hygiene — The main aim of sleep hygiene education is to provide participants with a set of behavioral and environmental recommendations intended to promote healthy sleep. During the intervention, participants will become aware of their own sleep patterns, will learn about healthy sleep habits, and will be encouraged to follow a set of recommendations to improve their sleep. Key components of the intervention are sleep hygiene and education.

SUMMARY:
The overall goal of this project is to evaluate the effect of enhanced psychological well-being on sleep quality. This study will demonstrate whether combining an intervention designed to promote psychological well-being with sleep hygiene education improves sleep quality in a non-clinical population of distressed adults reporting poor sleep in the absence of a diagnosed sleep disorder. The investigators expect an intervention combining elements of psychological well-being and sleep hygiene education to result in significant improvements in sleep quality measures from baseline to post-intervention, and greater improvements in sleep quality measures at post-intervention as compared with sleep hygiene education alone.

DETAILED DESCRIPTION:
Psychological distress is often associated with poor sleep quality. The role of psychological well-being has often been neglected and most interventions for sleep improvement have focused primarily on sleep disorders. This approach is limited to those individuals who have specific conditions and little resources have been directed to the promotion of sleep quality in the general population.

This study will be a pilot parallel-arm, randomized controlled trial to assess the baseline associations between psychological well-being and different measures of sleep outcomes, determine the effect of elements of a psychological well-being promoting intervention on sleep quality, and examine effect size estimates of key sleep-related outcomes (duration, efficiency, quality) to provide essential data to inform a main efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Distress according to the Perceived Stress Scale
* Poor sleep quality according to the Pittsburgh Sleep Quality Index
* No diagnosis of sleep disorders
* English fluency
* Access to a computer with an Internet connection

Exclusion Criteria:

* Inability to provide informed consent for any reason
* Cognitive impairment according to the Montreal Cognitive Assessment
* Suspected presence of sleep apnea according to the Berlin Questionnaire
* Diagnosis of a chronic medical or psychiatric condition
* Severe depression or suicidal thoughts or wishes according to the Beck Depression Inventory
* Body Mass Index (BMI) ≥ 35 kg/m2
* Chronic use of medications for sleep or chronic medical and psychiatric conditions
* Any current psychological or behavioral intervention administered by a health care provider or as part of a research project
* Shift workers
* Pregnant women
* Parents or caregivers of newborns (<1 year)
* Heavy drinkers (≥ 8 drinks/week for women and ≥ 15 drinks/week for men)
* Binge drinkers (≥ 4 drinks on a single occasion within about 2 hours for women and ≥ 5 drinks on a single occasion within about 2 hours for men
* Use of recreational or street drugs
* Heavy smokers (≥ 20 cigarettes daily)
* Heavy caffeine users (> 400 mg a day, corresponding to about 4 or 5 cups of coffee)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality: Pittsburgh Sleep Quality Index (PSQI) | Baseline to immediate post-intervention
  Measured by the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-rating scale for the assessment of sleep quality over a 1-month time interval. The PSQI yields 7 component scores and one global score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is given a score from 0-3. The global score is calculated by summing the seven component scores, providing an overall score ranging from 0-21, where lower scores indicate a higher sleep quality.
Change in insomnia severity: Insomnia Severity Index (ISI) | Baseline to immediate post-intervention
  Measured by the Insomnia Severity Index (ISI), a 7-item self-rated questionnaire to measure insomnia severity in the past 2 weeks. The total score ranges from 0-28, with higher scores indicating greater severity of insomnia. Scores of 8-14, 15-21, and 22-28 are indicative of subthreshold, moderate, and severe clinical insomnia, respectively.
Changes in total sleep time | Baseline to immediate post-intervention
  Measured by self-reported sleep diary
Changes in sleep onset latency | Baseline to immediate post-intervention
  Measured by self-reported sleep diary
Changes in wake after sleep onset | Baseline to immediate post-intervention
  Measured by self-reported sleep diary

SECONDARY OUTCOMES:
Change in psychological distress | Baseline to immediate post-intervention
  Measured by the Symptom Questionnaire (SQ), a 92-item self-rating scale for the assessment of psychological distress over a 1-week time interval. The SQ yields 4 main scales: anxiety, depression, somatization, and hostility. Each scale can be further divided into 2 sub-scales: one concerned with symptoms (17 items) and the other with well-being (6 items). Answers on each item are dichotomous (i.e., yes/no or true false). Scales and subscales can be scored separately, and the sum of the 4 main scale scores yields a total distress score. A response of yes/true for a symptom item gives 1 point, and a response of no/false for a well-being question gives 1 point for a score ranging from 0-23 for each main scale and 0-17 for each subscale, where a higher score indicates greater distress. If the well-being score is calculated separately the raw score can be subtracted from 6 for a score ranging from 0-6, where a higher score indicates greater well-being.
Change in psychological well-being | Baseline to immediate post-intervention
  Measured by the Psychological Well-being scale, a 42-item self-rating scale for the assessment of 6 dimensions of psychological well-being: self-acceptance, positive relations with others, autonomy, environmental mastery, purpose in life, and personal growth. Each of the 42 six-point response items are given a score from 1-6, with questions phrased in the negative reversed (e.g., 1 to 6, 6 to 1). The total score in each dimension ranges from 7-42, and all the dimensions scores are summed to give a final total ranging from 42-252, with higher scores indicating greater psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators can request de-identified data after the primary outcomes of this research project are published. Requests should be made in writing to the PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after the completion of the study.
Access Criteria: Request data in writing by contacting the PI.

REFERENCES:
- [Background] Almojali AI, Almalki SA, Alothman AS, Masuadi EM, Alaqeel MK. The prevalence and association of stress with sleep quality among medical students. J Epidemiol Glob Health. 2017 Sep;7(3):169-174. doi: 10.1016/j.jegh.2017.04.005. Epub 2017 May 5. PMID 28756825
- [Background] Bao YP, Han Y, Ma J, Wang RJ, Shi L, Wang TY, He J, Yue JL, Shi J, Tang XD, Lu L. Cooccurrence and bidirectional prediction of sleep disturbances and depression in older adults: Meta-analysis and systematic review. Neurosci Biobehav Rev. 2017 Apr;75:257-273. doi: 10.1016/j.neubiorev.2017.01.032. Epub 2017 Feb 6. PMID 28179129
- [Background] Bermudez-Millan A, Perez-Escamilla R, Segura-Perez S, Damio G, Chhabra J, Osborn CY, Wagner J. Psychological Distress Mediates the Association between Food Insecurity and Suboptimal Sleep Quality in Latinos with Type 2 Diabetes Mellitus. J Nutr. 2016 Oct;146(10):2051-2057. doi: 10.3945/jn.116.231365. Epub 2016 Aug 3. PMID 27489004
- [Background] Benasi G, Guidi J, Rafanelli C, Fava GA. New applications of Well-Being Therapy. Rivista Sperimentale di Freniatria, 1:87-106, 2019
- [Background] Buysse DJ. Sleep health: can we define it? Does it matter? Sleep. 2014 Jan 1;37(1):9-17. doi: 10.5665/sleep.3298. PMID 24470692
- [Background] Chida Y, Steptoe A. Positive psychological well-being and mortality: a quantitative review of prospective observational studies. Psychosom Med. 2008 Sep;70(7):741-56. doi: 10.1097/PSY.0b013e31818105ba. Epub 2008 Aug 25. PMID 18725425
- [Background] Czeisler CA. Impact of sleepiness and sleep deficiency on public health--utility of biomarkers. J Clin Sleep Med. 2011 Oct 15;7(5 Suppl):S6-8. doi: 10.5664/JCSM.1340. PMID 22003334
- [Background] Fava GA, Sonino N. Psychosomatic assessment. Psychother Psychosom. 2009;78(6):333-41. doi: 10.1159/000235736. Epub 2009 Aug 27. PMID 19713727
- [Background] Fava GA. Well-Being Therapy treatment manual and clinical applications. Basel: Karger, 2016.
- [Background] Fava GA. Well-Being Therapy: Current Indications and Emerging Perspectives. Psychother Psychosom. 2016;85(3):136-45. doi: 10.1159/000444114. Epub 2016 Apr 5. No abstract available. PMID 27043240
- [Background] Franzen PL, Buysse DJ. Sleep disturbances and depression: risk relationships for subsequent depression and therapeutic implications. Dialogues Clin Neurosci. 2008;10(4):473-81. doi: 10.31887/DCNS.2008.10.4/plfranzen. PMID 19170404
- [Background] Irish LA, Kline CE, Gunn HE, Buysse DJ, Hall MH. The role of sleep hygiene in promoting public health: A review of empirical evidence. Sleep Med Rev. 2015 Aug;22:23-36. doi: 10.1016/j.smrv.2014.10.001. Epub 2014 Oct 16. PMID 25454674
- [Background] Jahoda M. Current concepts of positive mental health. New York, NY, US: Basic Books, 1958.
- [Background] Leger D, Poursain B, Neubauer D, Uchiyama M. An international survey of sleeping problems in the general population. Curr Med Res Opin. 2008 Jan;24(1):307-17. doi: 10.1185/030079907x253771. PMID 18070379
- [Background] Lund HG, Reider BD, Whiting AB, Prichard JR. Sleep patterns and predictors of disturbed sleep in a large population of college students. J Adolesc Health. 2010 Feb;46(2):124-32. doi: 10.1016/j.jadohealth.2009.06.016. Epub 2009 Aug 3. PMID 20113918
- [Background] Murawski B, Wade L, Plotnikoff RC, Lubans DR, Duncan MJ. A systematic review and meta-analysis of cognitive and behavioral interventions to improve sleep health in adults without sleep disorders. Sleep Med Rev. 2018 Aug;40:160-169. doi: 10.1016/j.smrv.2017.12.003. Epub 2017 Dec 29. PMID 29397329
- [Background] Ohayon MM. Epidemiology of insomnia: what we know and what we still need to learn. Sleep Med Rev. 2002 Apr;6(2):97-111. doi: 10.1053/smrv.2002.0186. PMID 12531146
- [Background] Ohayon MM, O'Hara R, Vitiello MV. Epidemiology of restless legs syndrome: a synthesis of the literature. Sleep Med Rev. 2012 Aug;16(4):283-95. doi: 10.1016/j.smrv.2011.05.002. Epub 2011 Jul 26. PMID 21795081
- [Background] Pressman SD, Cohen S. Does positive affect influence health? Psychol Bull. 2005 Nov;131(6):925-971. doi: 10.1037/0033-2909.131.6.925. PMID 16351329
- [Background] Rafanelli C, Park SK, Ruini C, Ottolini F, Cazzaro M, Fava GA. Rating wellbeing and distress. Stress & Health 16(1): 55-61, 2000.
- [Background] Ryff CD. Psychological well-being revisited: advances in the science and practice of eudaimonia. Psychother Psychosom. 2014;83(1):10-28. doi: 10.1159/000353263. Epub 2013 Nov 19. PMID 24281296
- [Background] Seixas AA, Nunes JV, Airhihenbuwa CO, Williams NJ, Pandi-Perumal SR, James CC, Jean-Louis G. Linking emotional distress to unhealthy sleep duration: analysis of the 2009 National Health Interview Survey. Neuropsychiatr Dis Treat. 2015 Sep 25;11:2425-30. doi: 10.2147/NDT.S77909. eCollection 2015. PMID 26442563
- [Background] Scott D, Paterson JL, Happell B. Poor sleep quality in Australian adults with comorbid psychological distress and physical illness. Behav Sleep Med. 2014;12(4):331-41. doi: 10.1080/15402002.2013.819469. Epub 2013 Nov 1. PMID 24180418
- [Background] Tinetti ME, Bogardus ST Jr, Agostini JV. Potential pitfalls of disease-specific guidelines for patients with multiple conditions. N Engl J Med. 2004 Dec 30;351(27):2870-4. doi: 10.1056/NEJMsb042458. No abstract available. PMID 15625341
- [Background] Vaghela P, Sutin AR. Discrimination and sleep quality among older US adults: the mediating role of psychological distress. Sleep Health. 2016 Jun;2(2):100-108. doi: 10.1016/j.sleh.2016.02.003. Epub 2016 Apr 4. PMID 28923251
- [Background] Beck AT, Steer RA, Brown GK. Beck Depression Inventory: second edition manual. San Antonio (TX): The Psychological Corporation, 1996.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Fava GA, Guidi J. The pursuit of euthymia. World Psychiatry. 2020 Feb;19(1):40-50. doi: 10.1002/wps.20698. PMID 31922678
- [Background] Kellner R. A symptom questionnaire. J Clin Psychiatry. 1987 Jul;48(7):268-74. PMID 3597327
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Ryff CD. Happiness is everything or is it? Explorations on the meaning of psychological well-being. Journal of Personality and Social Psychology 57(6):1069-81, 1989.
- [Background] Spoormaker VI, Verbeek I, van den Bout J, Klip EC. Initial validation of the SLEEP-50 questionnaire. Behav Sleep Med. 2005;3(4):227-46. doi: 10.1207/s15402010bsm0304_4. PMID 16190812
- See also: American Academy of Sleep Medicine — http://sleepeducation.org/
- See also: National Sleep Foundation — http://www.sleepfoundation.org
- See also: National Institute of Health — https://www.nhlbi.nih.gov/health-topics/education-and-awareness/sleep-health